CLINICAL TRIAL: NCT06917768
Title: Oral Corticosteroids' Role in Pediatric Obstructive Sleep Apnea, a Non-Randomized Controlled Trial.
Brief Title: Oral Corticosteroids' Role in Pediatric Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hotel Dieu de France Hospital (Other)
Responsible Party: Principal Investigator, Oliver Majdalani, Principal Investigator, Hotel Dieu de France Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tfem/2023/50
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Obstructive Sleep Apnea
Keywords: Corticosteroids; Tonsillar hypertrophy; Pediatric OSA; Surgery; Coblation
MeSH Terms: interventions — Prednisolone

STUDY DESIGN:
Intervention Model Description: It is an interventional, prospective, non randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients undergoing surgical treatment (adenotonsillectomy). (Active Comparator): Children undergoing adenoidectomy and intracapsular tonsillectomy using Coblation™, by the same surgeon at HDF.
  Interventions: Procedure: Adenotonsillectomy
- Patients undergoing medical treatment (short-term and low dose oral corticosteroids). (Experimental): The second Group includes children whose parents have refused surgery despite informed understanding of the therapeutic algorithm of OSA. They received medical treatment consisting of a 1-month treatment with intranasal corticosteroids, coupled with a 5-day course of oral corticosteroids (prednisolone) at a safe dose of 1mg/kg.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Procedure: Adenotonsillectomy — Children undergoing adenoidectomy and intracapsular tonsillectomy using Coblation™, by the same surgeon at HDF.
  Other Names: Coblation
  Arms: Patients undergoing surgical treatment (adenotonsillectomy).
Drug: Prednisolone — The second Group includes children whose parents have refused surgery despite informed understanding of the therapeutic algorithm of OSA. They received medical treatment consisting of a 1-month treatment with intranasal corticosteroids, coupled with a 5-day course of oral corticosteroids (prednisolone) at a safe dose of 1mg/kg.
  Arms: Patients undergoing medical treatment (short-term and low dose oral corticosteroids).

SUMMARY:
This prospective interventional clinical trial (non-randomized) aims to evaluate oral corticosteroids' role as an alternative to surgery (gold-standard) in the treatment of obstructive sleep apnea in children. It also evaluates the evolution of symptoms' severity as well as any side effects linked to treatment.

This prospective study included children aged between 18 months and 8 years who consulted the same pediatric ENT physician's clinic for OSA secondary to adenotonsillar hypertrophy with no other comorbidities. They were divided into 2 Groups. Children undergoing intracapsular adenotonsillectomy by Coblation™ (Group 1) were compared to those receiving oral prednisolone at a dose of 1mg/kg for 5 days and 1 month of intranasal corticosteroids (Group 2). The follow-up tools were the Pediatric Sleep Questionnaire (PSQ) score and the size of the tonsils (Brodsky classification) evaluated at 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All children aged between 18 months and 8 years diagnosed with OSAS secondary to adenotonsillar hypertrophy

Exclusion Criteria:

* Children under 18 months or over 8 years old
* History of acute or chronic cardiorespiratory neuromuscular, or metabolic diseases
* Congenital craniofacial anomalies
* Chromosomal disorders
* Epilepsy

Ages: 18 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluate the effectiveness of low-dose, short-term oral corticosteroids in the treatment of OSA in children. | 6 months
  In Group 2, failure of medical treatment is defined by a persistence of apnea assessed by the clinician and parents and therefore a need for surgery within 6 months of follow-up, while therapeutic success reflects an improvement in symptoms and a disappearance of apnea documented by video, and therefore the absence of need for surgery after 6 months of follow-up.

SECONDARY OUTCOMES:
Evaluate the evolution of symptoms' severity | 6 months
  Evaluation at 1, 3 and 6 months of treatment (or surgery) the evolution of the OSA-related symptoms through the Pediatric Sleep Questionnaire.
  The Pediatric Sleep Questionnaire consists of 22 questions related to Pediatric OSA. The score is graded from 0 to 22 and is proportional to symptoms' severity (a higher score means a more severe sleep apnea).
Evaluate tonsils' size evolution with treatment | 6 months
  Evaluation at 1, 3 and 6 months of the evolution of tonsils' size through clinical evaluation using the Brodsky Score for tonsil size evaluation.
  Brodsky score can be 0, 1, 2, 3 or 4. A higher score reflects bigger tonsils.
Evaluate potential treatment-related side effects | 6 months
  Evaluation of any potential treatment-related side effect through clinical interrogation at 1,3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Rassi, Medical Doctor, Study Director — Hotel Dieu de France
Locations (1):
- Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fernandes RM, Wingert A, Vandermeer B, Featherstone R, Ali S, Plint AC, Stang AS, Rowe BH, Johnson DW, Allain D, Klassen TP, Hartling L. Safety of corticosteroids in young children with acute respiratory conditions: a systematic review and meta-analysis. BMJ Open. 2019 Aug 1;9(8):e028511. doi: 10.1136/bmjopen-2018-028511. PMID 31375615
- [Background] Mitchell RB, Pereira KD, Friedman NR. Sleep-disordered breathing in children: survey of current practice. Laryngoscope. 2006 Jun;116(6):956-8. doi: 10.1097/01.MLG.0000216413.22408.FD. PMID 16735907
- [Background] Meltzer LJ, Mindell JA. Sleep and sleep disorders in children and adolescents. Psychiatr Clin North Am. 2006 Dec;29(4):1059-76; abstract x. doi: 10.1016/j.psc.2006.08.004. PMID 17118282